CLINICAL TRIAL: NCT00666666
Title: A Phase II Study of AT101, to Abrogate BCL-2 Mediated Resistance to Androgen Ablation Therapy in Patients With Newly Diagnosed Stage D2 Prostate Cancer
Brief Title: R-(-)-Gossypol and Androgen Ablation Therapy in Treating Patients With Newly Diagnosed Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00264; 8014 (Other: NCI/CTEP); N01CM62201 (NIH); U01CA062491 (NIH); U01CA132194 (NIH); 080707 (Other: CINJ)
Record Dates: First submitted 2008-04-24; First posted 2008-04-25 (Estimated); Results first posted 2014-12-18 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-08

CONDITIONS: Adenocarcinoma of the Prostate; Stage IV Prostate Cancer
Keywords: prostate Cancer; adenocarcinoma of the prostate; stage IV prostate cancer; newly diagnosed stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gossypol acetic acid; bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AT101 (R-(-)-gossypol acetic acid) (Experimental): Patients will receive Hormone therapy with at least one LHRH agent (Leuprolide Acetate or Goserelin) for 6 weeks and include bicalutamide. Patients will begin AT101 daily at 6 weeks for 3 weeks of every 4 weeks (4 weeks - 1 cycle) and continue for 8 cycles of combined therapy (combined AT101, and LHRH agonist). After 8 cycles patients will continue hormonal therapy.
  Interventions: Drug: AT-101; Drug: Bicalutamide; Other: LHRH agent

INTERVENTIONS:
Drug: AT-101 — AT101 will be administered orally 20 mg/day for 21 days of a 28 day cycle.
  Other Names: R-(-)-gossypol acetic acid
Drug: Bicalutamide — Daily bicalutamide 50 mg po is encouraged for the first month of LHRH agonist therapy to prevent a flare. Continued bicalutamide use is optional. Bicalutamide will be administered orally at a dose of 50 mg po daily, Day 1 to 28 of each cycle.
  Other Names: Casodex; CDX
Other: LHRH agent — An LHRH agonist(Leuprolide Acetate or Goserelin)can be administered at standard dosing appropriate to the agent used.
  Other Names: Leutinizing Hormone Receptor Hormone agonist

SUMMARY:
This phase II trial is studying how well giving gossypol together with androgen ablation therapy works in treating patients with newly diagnosed metastatic prostate cancer. Gossypol may stop the growth of tumor cells by blocking blood flow to the tumor. Androgens can cause the growth of prostate tumor cells. Luteinizing hormone-releasing hormone agonists and drugs, such as bicalutamide, may lessen the amount of androgens made by the body. Giving gossypol together with androgen ablation therapy may be an effective treatment for prostate cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the percentage of patients with newly diagnosed metastatic prostate cancer who demonstrate undetectable prostate-specific antigen (PSA) (< 0.2 ng/mL) at 7 months when treated with R-(-)-gossypol (AT-101) and androgen ablation therapy.

SECONDARY OBJECTIVES:

I. To determine the safety of this regimen in these patients. II. To determine the percentage of patients with PSA >= 4.0 ng/mL, overall PSA < 4.0 ng/mL, and a PSA >= 0.2 ng/mL but < 4.0 ng/mL during the first 7 months of therapy.

OUTLINE:

Patients receive R-(-)-gossypol orally (PO) once daily (QD) on days 1-21. Treatment repeats every 28 weeks for 8 courses in the absence of disease progression or unacceptable toxicity. Patients may receive bicalutamide PO QD beginning 6 weeks before the initiation of R-(-)-gossypol and continuing after completion of treatment, at the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria

* Histologically proven adenocarcinoma of the prostate with clinical stage D2 disease defined by soft tissue or bony metastasis.
* Patients must have elevated PSA ≥ 5 ng/ml within 12 weeks prior to registration. Androgen ablation therapy, which must include an LHRH agonist, will begin 6 weeks prior to initiation of AT101.
* Patients are allowed prior local therapy with radiation or surgery. Patients must not have received more than 12 months of androgen ablation therapy or antiandrogen therapy in the adjuvant/neoadjuvant setting and no prior androgen ablation therapy for metastatic disease, beyond the six week induction period prior to initiation of AT101. Patients with prior adjuvant/neoadjuvant androgen ablation therapy must have completed such therapy at least 12 months prior.
* Must be 18 years old or older.
* Life expectancy of greater than 6 months.
* ECOG performance status ≤ 2.
* Patients must have normal organ and marrow function as defined below:

  * leukocytes ≥ 3,000/mcL
  * absolute neutrophil count ≥ 1,500/mcL
  * platelets ≥ 100,000/mcL
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 X institutional upper limit of normal
  * creatinine within normal institutional limits OR
  * creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* There must be no plans to receive concomitant chemotherapy or radiation therapy during the study period. Baseline and on study PSA values must be obtained from the same reference laboratory.
* The effects of AT101 on the developing human fetus at the recommended therapeutic dose are unknown. For this reason men and/or their partners must agree to use adequate contraception, (including hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation.

Exclusion Criteria

* Patients who have had radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients may not be receiving any other investigational agents.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to AT101 or other agents used in the study.
* Patients with bilateral orchiectomy are not eligible.
* Patients presenting with acute cord compression are not eligible.
* History of bowel obstruction or GI dismotility disorder.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow and retain AT-101 tablets.
* Requirement for routine use of hematopoietic growth factors (including granulocyte colony stimulating factor, granulocyte macrophage colony stimulating factor, or interleukin-11) or platelet transfusions to maintain absolute neutrophil counts or platelets counts above the required thresholds for study entry.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with AT-101.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-07; Primary Completion 2011-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert DiPaola, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (4):
- United States (4):
  - University of Chicago, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from April 2008 through July 2010, from four academic medical centers.
Pre-assignment Details: There are no pre-assignment requirements.
Groups:
- AT101 (R-(-)-Gossypol Acetic Acid): Patients will receive Hormone therapy with at least one LHRH agent (Leuprolide Acetate or Goserelin) for 6 weeks and include bicalutamide. Patients will begin AT101 daily at 6 weeks for 3 weeks of every 4 weeks (4 weeks - 1 cycle) and continue for 8 cycles of combined therapy (combined AT101, and LHRH agonist). After 8 cycles patients will continue hormonal therapy.
  AT-101 : AT101 will be administered orally 20 mg/day for 21 days of a 28 day cycle.
  Bicalutamide : Daily bicalutamide 50 mg po is encouraged for the first month of LHRH agonist therapy to prevent a flare. Continued bicalutamide use is optional. Bicalutamide will be administered orally at a dose of 50 mg po daily, Day 1 to 28 of each cycle.
  LHRH agent : An LHRH agonist(Leuprolide Acetate or Goserelin)can be administered at standard dosing appropriate to the agent used.
Period: Overall Study
Arm/Group | AT101 (R-(-)-Gossypol Acetic Acid)
Started | 55
Completed | 55
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | AT101 (R-(-)-Gossypol Acetic Acid)
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.58 (8.925)
Age, Continuous [Median (Full Range); unit: Years] | 61.5 [45 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 55
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 49
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 55
Gleason Score [Number; unit: participants] — A system of grading prostate cancer tissue based on how it looks under a microscope. Gleason scores range from 2 to 10 and indicate how likely it is that a tumor will spread. A low Gleason score means the cancer tissue is similar to normal prostate tissue and the tumor is less likely to spread; a high Gleason score means the cancer tissue is very different from normal and the tumor is more likely to spread.
  participants
    Gleason Score 6 | 1
    Gleason Score 7 | 13
    Gleason Score 8 | 12
    Gleason Score 9 | 24
    Gleason Score 10 | 3
    Not assessed | 2
Metastatic disease [Number; unit: participants]
  Visceral metastases | 3
  Bone/node metastases | 52

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Undetectable Prostate-specific Antigen (PSA) (< 0.2 ng/mL) at End of 7 Cycles
Time Frame: 3 years
Measure: Number; unit: percentage of participants
Arm/Group | AT101 (R-(-)-Gossypol Acetic Acid)
Number analyzed (Participants) | 55
percentage of participants | 22

2. Secondary Outcome: Percentage of Patients With PSA ≥ 0.2 ng/mL But < 4.0 ng/mL
Time Frame: 3 years
Measure: Number; unit: percentage of participants
Arm/Group | AT101 (R-(-)-Gossypol Acetic Acid)
Number analyzed (Participants) | 55
percentage of participants | 18

3. Secondary Outcome: Percentage of Patients With Overall PSA < 4.0 ng/mL
Time Frame: 3 years
Measure: Number; unit: percentage of participants
Arm/Group | AT101 (R-(-)-Gossypol Acetic Acid)
Number analyzed (Participants) | 55
percentage of participants | 60

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | AT101 (R-(-)-Gossypol Acetic Acid)
Serious Adverse Events (participants affected / at risk) | 13/55
Other Adverse Events (participants affected / at risk) | 55/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AT101 (R-(-)-Gossypol Acetic Acid) (N=55)
Eye disorders - optic neuritis (Eye disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 3 (3)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Infections and infestations - urosepsis (Infections and infestations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - left total hip arthroplasty (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AT101 (R-(-)-Gossypol Acetic Acid) (N=55)
Nausea (Gastrointestinal disorders) | 20 (28)
Vomiting (Gastrointestinal disorders) | 14 (22)
Constipation (Gastrointestinal disorders) | 13 (14)
Diarrhea (Gastrointestinal disorders) | 12 (18)
Abdominal pain (Gastrointestinal disorders) | 8 (11)
Flatulence (Gastrointestinal disorders) | 4 (4)
Fatigue (General disorders) | 32 (42)
Edema limbs (General disorders) | 5 (5)
Chills (General disorders) | 3 (3)
Pain (General disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 27 (42)
Anorexia (Metabolism and nutrition disorders) | 10 (12)
Hyperkalemia (Metabolism and nutrition disorders) | 8 (9)
Hypercalcemia (Metabolism and nutrition disorders) | 6 (10)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (7)
Acidosis (Metabolism and nutrition disorders) | 4 (5)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 19 (29)
Dizziness (Nervous system disorders) | 7 (8)
Headache (Nervous system disorders) | 6 (6)
Dysgeusia (Nervous system disorders) | 3 (3)
Peripheral motor neuropathy (Nervous system disorders) | 3 (4)
Alanine aminotransferase increased (Investigations) | 23 (35)
Aspartate aminotransferase increased (Investigations) | 17 (26)
Creatinine increased (Investigations) | 10 (17)
Platelet count decreased (Investigations) | 6 (15)
Alkaline phosphatase increased (Investigations) | 5 (6)
White blood cell decreased (Investigations) | 5 (12)
Lymphocyte count decreased (Investigations) | 3 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (10)
Bone pain (Musculoskeletal and connective tissue disorders) | 7 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 22 (34)
Hot flashes (Vascular disorders) | 19 (22)
Hypertension (Vascular disorders) | 6 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (8)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (4)
Urinary frequency (Renal and urinary disorders) | 8 (8)
Urinary tract pain (Renal and urinary disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 6 (6)
Depression (Psychiatric disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Erectile dysfunction (Reproductive system and breast disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less